CLINICAL TRIAL: NCT02734004
Title: A Phase I/II Study of MEDI4736 (Anti-PD-L1 Antibody) in Combination With Olaparib (PARP Inhibitor) in Patients With Advanced Solid Tumors
Brief Title: A Phase I/II Study of MEDI4736 in Combination With Olaparib in Patients With Advanced Solid Tumors.
Acronym: MEDIOLA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D081KC00001; 2015-004005-16 (EudraCT Number)
Expanded Access: NCT03079687 (Approved for marketing)
Record Dates: First submitted 2016-03-17; First posted 2016-04-12 (Estimated); Results first posted 2023-10-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ovarian; Breast; SCLC; Gastric Cancers
Keywords: MEDIOLA; Olaparib; MEDI4736; Bevacizumab; Ovarian cancer; Breast cancer; Small Cell Lung Cancer; Gastric Cancer; Phase I/II, Adults; PDL-1
MeSH Terms: conditions — Stomach Neoplasms; Ovarian Neoplasms; Breast Neoplasms; Small Cell Lung Carcinoma | interventions — olaparib; durvalumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Includes initial stage cohorts (modules 1 to 4): Olaparib twice daily starting on week 1 day 1 and MEDI4736 every 4 weeks starting on week 5 day 1
  Interventions: Drug: Olaparib; Drug: MEDI4736
- Arm 2 (Experimental): Includes 2nd stage cohorts (modules 5 & 7): Olaparib twice daily starting on week 1 day 1 and MEDI4736 every 4 weeks starting on week 1 day 1
  Interventions: Drug: Olaparib; Drug: MEDI4736
- Arm 3 (Experimental): Includes 2nd stage cohort (module 6): Olaparib twice daily starting on week 1 day 1 / MEDI4736 every 4 weeks starting on week 1 day 1 / Bevacizumab every 2 weeks starting on week 1 day 1
  Interventions: Drug: Olaparib; Drug: MEDI4736; Drug: Bevacizumab

INTERVENTIONS:
Drug: Olaparib — Olaparib
Drug: MEDI4736 — MEDI4736
Drug: Bevacizumab — Bevacizumab
  Other Names: Avastin
  Arms: Arm 3

SUMMARY:
The purpose of this study is to look at the effectiveness, safety, and antitumor activity of study drugs MEDI4736 in combination with olaparib (modules 1, 2, 3, 4, 5 and 7) and MEDI4736 in combination with olaparib and bevacizumab (module 6). It will also examine what happens to the study drugs in the body and investigate how well the combination between MEDI4736, olaparib and bevacizumab is tolerated.

DETAILED DESCRIPTION:
This is a phase I/II open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK) and antitumor activity of MEDI4736 in combination with olaparib in patients with advanced solid tumors, selected based on a rationale for response to olaparib.

Patients will be poly (adenosine diphosphate-ribose) polymerase (PARP)-inhibitor and immunotherapy (IMT)-naïve (defined as no prior exposure to PARP inhibitors or IMT, including, but not limited to, other anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], anti-programmed cell death 1 [PD-1], anti-programmed death-ligand 1 [PD-L1] monoclonal antibodies, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).

The 4 initial stage cohorts (Modules 1 to 4) include patients with relapsed small cell lung cancer (SCLC), germline BRCA mutated (gBRCAm) metastatic human epidermal growth factor receptor 2 (HER2)-negative breast cancer, gBRCAm platinum-sensitive relapsed ovarian cancer, and gastric cancer. The data cut-off occurred once all 4 Modules had reached last patient first visit (LPFV) + 2 years and all 4 cohorts had observed a median value for PFS.

Second stage cohorts (Modules 5 to 7) include patients with relapsed gBRCAm platinum-sensitive relapsed ovarian cancer and non gBRCAm platinum-sensitive relapsed ovarian cancer. The final data cut-off will be once Modules 6 and 7 have observed a median value for overall survival. At this timepoint, the clinical study database will close to new data.

ELIGIBILITY:
Inclusion criteria:

* Patients must have histologically or cytologically confirmed progressive advanced or metastatic solid tumor of one of the following:

  * Platinum sensitive relapsed small cell lung cancer (module 1)
  * gBRCAm HER2-negative metastatic breast cancer (module 2)
  * gBRCAm ovarian cancer (modules 3 and 5)
  * Metastatic or relapsed Gastric cancer (adenocarcinoma) (module 4)
  * gBRCAm negative ovarian cancer (modules 6 and 7)
* At least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) (or magnetic resonance imaging [MRI] suitable for assessment as per RECIST 1.1. The baseline scan must be obtained within 28 days prior to the first dose of olaparib.
* Male or female patients, age ≥18 years (≥19 years for South Korea)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy ≥12 weeks
* Adequate organ and marrow function
* Ability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation. Patients should not have gastrointestinal illnesses that would preclude the absorption of olaparib, which is an oral agent. For the gastric cancer cohort, patients with a full or partial gastrectomy will be permitted.
* Ability of patient to understand and the willingness to sign a written informed consent document prior to any protocol related procedures, including screening evaluations.
* Female patients must either:

  * Be of non-reproductive potential OR
  * Have a negative serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on Day 1, and agree to use contraception if they or their partner are of reproductive potential

Exclusion criteria

* Prior chemotherapy or other systemic anticancer therapy within 4 weeks prior to start of olaparib treatment, 6 weeks for nitrosoureas or mitomycin. Exceptions include: Anti-hormonal treatment for ER positive or PR positive breast cancer is allowed until 7 days prior to treatment with olaparib, exposure to an investigational agent within 30 days or 5 half-lives (whichever is the longer) prior to start of olaparib treatment is not allowed, prior receipt of biologics targeting T cell co-regulatory proteins and/or immune checkpoints is not allowed. Examples include MEDI4736 or other PD1 or PD-L1 or PD-L2 inhibitors or anti-CTLA4 therapy, previous treatment with a PARP inhibitor, is not allowed.
* Radiation therapy within 4 weeks prior to start of olaparib treatment (includes radiation targeting bone metastases) or radionuclide treatment within 6 weeks of treatment start.
* Current dependency on total parenteral nutrition or IV fluid hydration.
* Concomitant use of known strong cytochrome P450 (CYP) 3A (CYP3A) inhibitors or moderate CYP3A inhibitors. Concomitant use of known strong or moderate CYP3A inducers.
* Concomitant therapy with any other anticancer therapy or chronic use of systemic corticosteroids.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation
* Whole blood transfusions in the last 120 days
* Patients with symptomatic or uncontrolled brain metastases.
* Patients being considered at poor medical risk due to a serious, uncontrolled medical disorder or non-malignant systemic disease.
* Any psychiatric disorder that prohibits obtaining informed consent
* Major surgery or significant traumatic injury within 2 weeks of run-in
* Immunocompromised patients
* QTc prolongation >470 msec or other significant ECG abnormality noted within 14 days of treatment
* Pregnant and breastfeeding women are excluded.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrolment in the present study
* Participation in a clinical study within 28 days or 5 half-lives of the drug, whichever is longer.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2026-09-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Domchek, MD, Principal Investigator — Abramson Cancer Center, University of Pennsylvania
Locations (40):
- United States (7):
  - Research Site, Newnan, Georgia
  - Research Site, Towson, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Hilliard, Ohio
  - Research Site, Philadelphia, Pennsylvania
- France (10):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Dijon
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pierre Benit Cedex
  - Research Site, Toulouse
  - Research Site, Villejuif
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Netherlands (5):
  - Research Site, Amsterdam
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Utrecht
- South Korea (3):
  - Research Site, Goyang-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Switzerland (2):
  - Research Site, Chur
  - Research Site, Lausanne
- United Kingdom (8):
  - Research Site, Cambridge
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Greater London
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Sutton

REFERENCES:
- [Derived] Drew Y, Kim JW, Penson RT, O'Malley DM, Parkinson C, Roxburgh P, Plummer R, Im SA, Imbimbo M, Ferguson M, Rosengarten O, Steeghs N, Kim MH, Gal-Yam E, Tsoref D, Kim JH, You B, De Jonge M, Lalisang R, Gort E, Bastian S, Meyer K, Feeney L, Baker N, Ah-See ML, Domchek SM, Banerjee S; MEDIOLA Investigators. Olaparib plus Durvalumab, with or without Bevacizumab, as Treatment in PARP Inhibitor-Naive Platinum-Sensitive Relapsed Ovarian Cancer: A Phase II Multi-Cohort Study. Clin Cancer Res. 2024 Jan 5;30(1):50-62. doi: 10.1158/1078-0432.CCR-23-2249. PMID 37939124
- [Derived] Staniszewska AD, Armenia J, King M, Michaloglou C, Reddy A, Singh M, San Martin M, Prickett L, Wilson Z, Proia T, Russell D, Thomas M, Delpuech O, O'Connor MJ, Leo E, Angell H, Valge-Archer V. PARP inhibition is a modulator of anti-tumor immune response in BRCA-deficient tumors. Oncoimmunology. 2022 Jun 18;11(1):2083755. doi: 10.1080/2162402X.2022.2083755. eCollection 2022. PMID 35756843
- [Derived] Domchek SM, Postel-Vinay S, Im SA, Park YH, Delord JP, Italiano A, Alexandre J, You B, Bastian S, Krebs MG, Wang D, Waqar SN, Lanasa M, Rhee J, Gao H, Rocher-Ros V, Jones EV, Gulati S, Coenen-Stass A, Kozarewa I, Lai Z, Angell HK, Opincar L, Herbolsheimer P, Kaufman B. Olaparib and durvalumab in patients with germline BRCA-mutated metastatic breast cancer (MEDIOLA): an open-label, multicentre, phase 1/2, basket study. Lancet Oncol. 2020 Sep;21(9):1155-1164. doi: 10.1016/S1470-2045(20)30324-7. Epub 2020 Aug 6. PMID 32771088
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081KC00001&attachmentIdentifier=54f68400-a701-4a0d-8cab-0b0cc000d3c4&fileName=D081KC00001_CSP-v7_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081KC00001&attachmentIdentifier=ceade008-aa3e-4dea-8e71-4e0eb7db1cc5&fileName=D081KC00001_CSR_Synopsis_Redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081KC00001&attachmentIdentifier=d52a57f7-cf47-4fc2-ba93-9357db074c41&fileName=D081KC00001_SAP_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase I/II open-label study was conducted in participants with advanced solid tumors at 43 centers in France, the United Kingdom, the Republic of Korea, the USA, the Netherlands, Israel, and Switzerland. Initial stage cohorts: Results are reported for analysis with assessment until data cut-off (DCO) of 14 Jun 2019 [except for overall survival (OS) for ovarian cancer cohort (DCO: 17 Sep 2021)]. Second stage cohorts: Results are reported for analysis with assessment until DCO of 17 Sep 2021.
Pre-assignment Details: This study consists a screening period (28 days), run-in monotherapy treatment period (initial stage cohort only; 4 weeks) followed by combination therapy treatment period until progressive disease (PD). 148 participants entered initial stage cohorts and 114 participants entered second stage cohorts. Thus, 262 participants were enrolled in the study.
Groups:
- Initial Stage: Small Cell Lung Cancer: Participants received monotherapy with olaparib 300 milligram (mg) orally twice daily for 4 weeks. Participants then continued to receive combination therapy with olaparib and MEDI4736 1.5 grams (g) intravenous (IV) infusion every 4 weeks in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Initial Stage: Breast Cancer; Initial Stage: Ovarian Cancer; Initial Stage: Gastric Cancer: Participants received monotherapy with olaparib 300 mg orally twice daily for 4 weeks. Participants then continued to receive combination therapy with olaparib and MEDI4736 1.5 g IV infusion every 4 weeks in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Second Stage: Ovarian Cancer Expansion; Second Stage: Ovarian Cancer Doublet: Participants received combination therapy with olaparib 300 mg orally twice daily and MEDI4736 1.5 g IV infusion every 4 weeks in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Second Stage: Ovarian Cancer Triplet: Participants received combination therapy with olaparib 300 mg orally twice daily plus MEDI4736 1.5 g IV infusion every 4 weeks plus bevacizumab 10 mg/kilogram (kg) IV infusion every 2 weeks in 28-day cycle until PD or specific treatment discontinuation criteria were met.
Period: Overall Study
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Started | 40 | 34 | 34 | 40 | 51 | 31 | 32
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 40 | 34 | 34 | 40 | 51 | 31 | 32
Not completed — Death | 36 | 24 | 26 | 35 | 13 | 17 | 20
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1 | 3 | 0 | 2
Not completed — Other | 0 | 8 | 7 | 4 | 34 | 14 | 10

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least 1 dose of study treatment and had no important protocol deviation resulting in exclusion from the analysis set as defined in the Statistical Analysis Plan (i.e, not meeting key eligibility criteria).
Groups:
- Initial Stage: Small Cell Lung Cancer; Initial Stage: Breast Cancer; Initial Stage: Ovarian Cancer; Initial Stage: Gastric Cancer: Participants received monotherapy with olaparib 300 mg orally twice daily for 4 weeks. Participants then continued to receive combination therapy with olaparib and MEDI4736 1.5 g IV infusion every 4 weeks in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Second Stage: Ovarian Cancer Triplet: Participants received combination therapy with olaparib 300 mg orally twice daily plus MEDI4736 1.5 g IV infusion every 4 weeks plus bevacizumab 10 mg/kg IV infusion every 2 weeks in 28-day cycle until PD or specific treatment discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet | Total
Number analyzed (Participants) | 38 | 30 | 32 | 39 | 51 | 31 | 32 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 29 | 27 | 29 | 38 | 17 | 12 | 175
  >=65 years | 15 | 1 | 5 | 10 | 13 | 14 | 20 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 29 | 32 | 13 | 51 | 31 | 32 | 205
  Male | 21 | 1 | 0 | 26 | 0 | 0 | 0 | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 17 | 22 | 24 | 34 | 20 | 24 | 162
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 6 | 7 | 6 | 13 | 12 | 10 | 3 | 57
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Missing | 11 | 6 | 4 | 2 | 4 | 0 | 5 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 24 | 28 | 37 | 47 | 30 | 27 | 220
  Missing | 11 | 6 | 4 | 2 | 4 | 0 | 5 | 32

OUTCOME MEASURES:

1. Primary Outcome: Initial Stage Cohorts: Disease Control Rate (DCR) at Week 12
Description: The DCR at 12 weeks was defined as the percentage of participants who had complete response (CR) + partial response (PR) + stable disease (SD) at 12 weeks. Participants demonstrated SD for a minimum interval of 11 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e. 77 days) following the start of treatment. The DCR was determined using Investigator assessments according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Time Frame: RECIST performed at baseline, at 4 weeks after first dose of olaparib monotherapy and every 8 weeks +/-7 days thereafter. Assessed until DCO 14 Jun 2019.
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer
Number analyzed (Participants) | 38 | 30 | 32 | 39
percentage of participants | 28.9 | 80.0 | 81.3 | 25.6

2. Primary Outcome: Second Stage Cohort: Objective Response Rate (ORR)
Description: The ORR (based on RECIST 1.1 as assessed by the Investigator) was defined as the percentage of participants with at least 1 visit response of CR or PR prior to PD or last evaluable assessment in the absence of progression. The 95% confidence interval (CI) were calculated using Exact Clopper-Pearson confidence limits for the binomial proportion.
Time Frame: RECIST performed at baseline, and every 8 weeks +/-7 days thereafter. Assessed until 17 Sep 2021.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Second Stage: Ovarian Cancer Expansion
Number analyzed (Participants) | 51
percentage of participants | 92.2 [81.12 to 97.82]

3. Primary Outcome: Second Stage Cohorts: DCR at Week 24
Description: The DCR at 24 weeks was defined as the percentage of participants who had CR + PR + SD at 24 weeks. Participants demonstrated SD for a minimum interval of 23 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e. 161 days) following the start of treatment. The DCR was determined using Investigator assessments according to RECIST v1.1.
Time Frame: RECIST performed at baseline, and every 8 weeks +/-7 days thereafter. Assessed until 17 Sep 2021.
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 31 | 32
percentage of participants | 74.2 | 28.1

4. Secondary Outcome: Second Stage Expansion Cohort: DCR at Week 24
Description: as for outcome 3
Time Frame: RECIST performed at baseline, and every 8 weeks +/-7 days thereafter. Assessed until 17 Sep 2021.
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Second Stage: Ovarian Cancer Expansion
Number analyzed (Participants) | 51
percentage of participants | 88.2

5. Secondary Outcome: Initial Stage Cohorts: DCR at Week 28
Description: The DCR at 28 weeks was defined as the percentage of participants who had CR + PR + SD at 28 weeks. Participants demonstrated SD for a minimum interval of 27 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e. 189 days) following the start of treatment. The DCR was determined using Investigator assessments according to RECIST v1.1.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer
Number analyzed (Participants) | 38 | 30 | 32 | 39
percentage of participants | 5.3 | 50.0 | 65.6 | 7.7

6. Secondary Outcome: Second Stage Cohorts: DCR at Week 56
Description: The DCR at 56 weeks was defined as the percentage of participants who had CR + PR + SD at 56 weeks. Participants demonstrated SD for a minimum interval of 55 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e. 385 days) following the start of treatment. The DCR was determined using Investigator assessments according to RECIST v1.1.
Time Frame: RECIST performed at baseline, and every 8 weeks +/-7 days thereafter. Assessed until 17 Sep 2021.
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 51 | 31 | 32
percentage of participants | 41.2 | 38.7 | 9.4

7. Secondary Outcome: Initial and Second Stage Cohorts: ORR
Description: The ORR (based on RECIST 1.1 as assessed by the Investigator) was defined as the percentage of participants with at least 1 visit response of CR or PR prior to PD or last evaluable assessment in the absence of progression. The 95% CI were calculated using Exact Clopper-Pearson confidence limits for the binomial proportion.
Time Frame: RECIST performed at baseline, at 4 weeks after first dose of olaparib monotherapy (for initial stage cohort only) and every 8 weeks +/-7 days thereafter. Assessed until DCO 14 Jun 2019 and 17 Sep 2021 for initial and second stage cohorts, respectively
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 38 | 30 | 32 | 39 | 31 | 32
percentage of participants | 10.5 [2.94 to 24.80] | 63.3 [43.86 to 80.07] | 71.9 [53.25 to 86.25] | 10.3 [2.87 to 24.22] | 87.1 [70.17 to 96.37] | 34.4 [18.57 to 53.19]

8. Secondary Outcome: Initial and Second Stage Cohorts: Duration of Response (DoR)
Description: The DoR (based on RECIST 1.1 as assessed by the Investigator) was defined as the time from the date of first documented response until date of documented progression or death in the absence of PD. The DoR was calculated using Kaplan-Meier technique.
Time Frame: as for outcome 7
Population: The full analysis set included all participants who received at least 1 dose of study treatment and had no important protocol deviation resulting in exclusion from the analysis set as defined in the Statistical Analysis Plan (i.e, not meeting key eligibility criteria). Only participants with objective response were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 4 | 19 | 23 | 4 | 47 | 27 | 11
months | 3.6 [2.6 to 4.6] | 9.2 [5.5 to 20.3] | 10.2 [5.7 to 22.3] | 14.8 [6.4 to NA] — Upper limit of Inter-quartile range was not reached. | 14.8 [9.0 to NA] — Upper limit of Inter-quartile range was not reached. | 11.1 [7.4 to 22.1] | 6.9 [5.4 to 11.1]

9. Secondary Outcome: Initial and Second Stage Cohorts: Progression-Free Survival (PFS)
Description: The PFS (based on RECIST 1.1 as assessed by the Investigator) was defined as the time from start of study treatment (Day 1; start of olaparib monotherapy for initial stage cohorts) until the date of objective PD or death (by any cause in the absence of disease progression) regardless of whether the patient withdraws from therapy or receives another anticancer therapy prior to disease progression. The PFS was calculated using Kaplan-Meier technique.
Time Frame: as for outcome 7
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 38 | 30 | 32 | 39 | 51 | 31 | 32
months | 2.4 [0.9 to 3.0] | 8.2 [4.6 to 11.8] | 12.0 [8.2 to 15.9] | 2.6 [1.4 to 2.8] | 15.0 [12.9 to 24.1] | 14.7 [9.2 to 18.1] | 5.5 [3.6 to 7.5]

10. Secondary Outcome: Initial Stage Cohorts: Percentage Change From Baseline in Target Tumor Size at Weeks 12 and 28
Description: The percentage change in target tumor size at each timepoint (based on RECIST 1.1 target lesion measurements) was obtained for each participant taking the difference between the sum of the target lesions at each timepoint and the sum of the target lesions at baseline divided by the sum of the target lesions at baseline times 100. Baseline was defined as the last evaluable assessment prior to starting olaparib treatment.
Time Frame: Baseline (Day 1) and Weeks 12 and 28. Assessed until DCO 14 Jun 2019
Population: The full analysis set included all participants who received at least 1 dose of study treatment and had no important protocol deviation resulting in exclusion from the analysis set as defined in the Statistical Analysis Plan (i.e, not meeting key eligibility criteria). Only participants with either a tumor size recorded at 12 and 28 weeks or enough information to impute a value were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in tumor size
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer
Number analyzed (Participants) | 22 | 29 | 29 | 21
percentage change in tumor size
  Week 12 | 17.23 (54.752) | -26.13 (43.033) | -35.86 (29.791) | 20.81 (75.944)
  Week 28: number analyzed (Participants) | 5 | 19 | 26 | 4
  Week 28 | -2.05 (15.671) | -40.85 (39.541) | -53.74 (31.147) | -41.00 (43.625)

11. Secondary Outcome: Second Stage Cohorts: Percentage Change From Baseline in Target Tumor Size at Weeks 24 and 56
Description: The percentage change in target tumor size at each timepoint (based on RECIST 1.1 target lesion measurements) was obtained for each participant taking the difference between the sum of the target lesions at each timepoint and the sum of the target lesions at baseline divided by the sum of the target lesions at baseline times 100. Baseline was defined as the last assessment prior to Cycle 1 Day 1.
Time Frame: Baseline (Day 1) and Weeks 24 and 56. Assessed until DCO 17 Sep 2021
Population: The full analysis set included all participants who received at least 1 dose of study treatment and had no important protocol deviation resulting in exclusion from the analysis set as defined in the Statistical Analysis Plan (i.e, not meeting key eligibility criteria). Only participants with either a tumor size recorded at 24 and 56 weeks or enough information to impute a value were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in tumor size
Arm/Group | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 47 | 27 | 15
percentage change in tumor size
  Week 24 | -66.30 (26.672) | -43.00 (32.432) | -35.63 (34.001)
  Week 56: number analyzed (Participants) | 26 | 15 | 5
  Week 56 | -77.74 (26.472) | -60.00 (29.058) | -39.54 (33.719)

12. Secondary Outcome: Initial and Second Stage Cohorts: Best Percentage Change From Baseline in Target Tumor Size
Description: The best percentage change from baseline in target tumor size was based on RECIST 1.1 target lesion measurements taken at each RECIST 1.1 assessment. All measurements until PD or the last evaluable assessment in the absence of PD was included in the calculation. Baseline was defined as the last evaluable assessment prior to starting olaparib treatment for initial stage cohorts. Baseline was defined as the last assessment prior to Cycle 1 Day 1 for second stage cohorts.
Time Frame: From baseline (Day 1) until confirmed PD/death. Assessed until DCO 14 Jun 2019 and 17 Sep 2021 for initial and second stage cohorts, respectively
Population: The full analysis set included all participants who received at least 1 dose of study treatment and had no important protocol deviation resulting in exclusion from the analysis set as defined in the Statistical Analysis Plan (i.e, not meeting key eligibility criteria). Only participants with at least 1 post baseline RECIST target lesion assessment scan were analyzed.
Measure: Mean (Standard Deviation); unit: percentage change in tumor size
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 36 | 30 | 31 | 37 | 51 | 31 | 32
percentage change in tumor size | 6.27 (32.398) | -47.60 (36.823) | -55.55 (35.789) | 1.64 (42.338) | -72.78 (31.497) | -53.30 (33.317) | -20.42 (41.160)

13. Secondary Outcome: Initial and Second Stage Cohorts: Time to Study Treatment Discontinuation or Death (TDT)
Description: The TDT was defined as the time from start of study treatment (Day 1; start of olaparib monotherapy for initial stage cohorts) to the earlier of the date of study treatment discontinuation or death. The TDT was calculated using the Kaplan-Meier technique.
Time Frame: From baseline (Day 1) until treatment discontinuation/death. Assessed until DCO 14 Jun 2019 and 17 Sep 2021 for initial and second stage cohorts, respectively
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 38 | 30 | 32 | 39 | 51 | 31 | 32
months | 2.8 [2.0 to 3.8] | 7.8 [6.2 to 12.1] | 13.1 [8.2 to 15.9] | 2.8 [2.1 to 3.2] | 19.3 [14.7 to 26.2] | 15.9 [10.3 to 18.4] | 6.6 [4.4 to 8.5]

14. Secondary Outcome: Initial and Second Stage Cohorts: OS
Description: The OS was defined as the time from the start of study treatment (Day 1; start of olaparib monotherapy for initial stage cohorts) until death due to any cause. The OS was calculated using the Kaplan-Meier technique.
Time Frame: From baseline (Day 1) until death from any cause. Assessed until DCO 14 Jun 2019 for initial stage cohorts except for ovarian cancer cohort and DCO 17 Sep 2021 for initial stage ovarian cancer cohort and second stage cohorts
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 38 | 30 | 32 | 39 | 51 | 31 | 32
months | 7.6 [5.6 to 8.8] | 20.5 [16.2 to 25.5] | 35.5 [27.2 to 50.7] | 6.4 [4.3 to 9.1] | NA [NA to NA] — Median and 95% CI had not reached. | 31.9 [22.1 to NA] — Upper limit of 95% CI had not reached. | 26.1 [18.7 to NA] — Upper limit of 95% CI had not reached.

15. Secondary Outcome: Initial and Second Stage Cohorts: Serum Concentrations of MEDI4736
Description: Blood samples were collected to determine the serum concentration of MEDI4736.
Time Frame: Pre-dose and within 10 minutes of end of infusion on Days 1, 85 and 113; Pre-dose on Days 29, 57 and 169; and 90 days post last dose of MEDI4736. Assessed until DCO 14 Jun 2019 and 17 Sep 2021 for initial and second stage cohorts, respectively
Population: The MEDI4736 pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of MEDI4736 and provided evaluable MEDI4736 PK profile for at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 36 | 34 | 32 | 36 | 51 | 31 | 32
microgram per milliliter (mcg/mL)
  Day 1: Pre-dose: number analyzed (Participants) | 36 | 33 | 32 | 36 | 42 | 30 | 31
  Day 1: Pre-dose | NA (NA) — NA = Below the lower limit of quantification (LLOQ). The LLOQ of MEDI4736 is 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of MEDI4736 is 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of MEDI4736 is 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of MEDI4736 is 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of MEDI4736 is 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of MEDI4736 is 0.05 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of MEDI4736 is 0.05 mcg/mL.
  Day 1: End of infusion: number analyzed (Participants) | 36 | 32 | 31 | 35 | 46 | 31 | 31
  Day 1: End of infusion | 483.5 (35.09) | 542.5 (36.04) | 417.9 (33.48) | 391.8 (25.09) | 409.3 (33.27) | 498.8 (30.27) | 397.1 (18.53)
  Day 29: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 43 | 31 | 31
  Day 29: Pre-dose |  |  |  |  | 93.56 (54.83) | 96.50 (34.67) | 78.23 (56.60)
  Day 57: Pre-dose: number analyzed (Participants) | 17 | 28 | 29 | 14 | 0 | 0 | 0
  Day 57: Pre-dose | 144.7 (38.96) | 165.2 (40.31) | 171.3 (31.73) | 114.7 (44.78) |  |  |
  Day 85: Pre-dose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 48 | 27 | 25
  Day 85: Pre-dose |  |  |  |  | 152.8 (50.14) | 145.2 (55.71) | 142.8 (63.07)
  Day 85: End of infusion: number analyzed (Participants) | 0 | 0 | 0 | 0 | 44 | 27 | 23
  Day 85: End of infusion |  |  |  |  | 610.6 (39.64) | 589.3 (35.48) | 482.9 (44.01)
  Day 113: Pre-dose: number analyzed (Participants) | 5 | 25 | 24 | 6 | 0 | 0 | 0
  Day 113: Pre-dose | 119.5 (44.27) | 220.7 (35.97) | 231.3 (33.45) | 196.9 (74.60) |  |  |
  Day 113: End of infusion: number analyzed (Participants) | 5 | 25 | 23 | 6 | 0 | 0 | 0
  Day 113: End of infusion | 504.8 (25.24) | 671.5 (31.79) | 585.5 (52.67) | 679.1 (34.80) |  |  |
  Day 169: Pre-dose: number analyzed (Participants) | 3 | 20 | 23 | 4 | 42 | 25 | 15
  Day 169: Pre-dose | 133.1 (30.74) | 231.5 (41.14) | 261.6 (45.92) | 230.7 (35.81) | 206.3 (61.24) | 162.6 (95.86) | 186.6 (65.36)
  90 days post last dose: number analyzed (Participants) | 3 | 6 | 8 | 6 | 8 | 9 | 9
  90 days post last dose | 6.907 (297.9) | 12.24 (4720) | 22.35 (120.9) | 17.23 (155.2) | 17.94 (331.8) | 17.47 (78.93) | 20.50 (340.0)

16. Secondary Outcome: Initial and Second Stage Cohorts: Serum Concentrations of Olaparib
Description: Blood samples were collected to determine the serum concentration of olaparib.
Time Frame: Pre-dose and 0.5-1 hour postdose on Days 1 and 22 of monotherapy; Pre-dose and 0.5-1, 1-3, 3-6 and 6-12 hours postdose on Day 15 of combination therapy. Assessed until DCO 14 Jun 2019 and 17 Sep 2021 for initial and second stage cohorts, respectively
Population: The olaparib PK analysis set included all participants who received at least 1 dose of olaparib and provided evaluable olaparib PK profile for at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 40 | 33 | 33 | 24 | 39 | 27 | 27
mcg/mL
  Monotherapy - Day 1: Pre-dose: number analyzed (Participants) | 40 | 31 | 33 | 24 | 0 | 0 | 0
  Monotherapy - Day 1: Pre-dose | NA (NA) — NA = Below LLOQ. The LLOQ of olaparib is 0.0005 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of olaparib is 0.0005 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of olaparib is 0.0005 mcg/mL. | NA (NA) — NA = Below LLOQ. The LLOQ of olaparib is 0.0005 mcg/mL. |  |  |
  Monotherapy - Day 1: 0.5-1 hour postdose: number analyzed (Participants) | 39 | 30 | 33 | 23 | 0 | 0 | 0
  Monotherapy - Day 1: 0.5-1 hour postdose | 3.647 (394.2) | 2.093 (1217) | 5.016 (150.1) | 2.321 (291.7) |  |  |
  Monotherapy - Day 22: Pre-dose: number analyzed (Participants) | 28 | 28 | 25 | 16 | 0 | 0 | 0
  Monotherapy - Day 22: Pre-dose | 1.374 (814.4) | 0.8500 (1501) | 1.242 (534.6) | 2.053 (124.6) |  |  |
  Monotherapy - Day 22: 0.5-1 hour postdose: number analyzed (Participants) | 26 | 25 | 26 | 17 | 0 | 0 | 0
  Monotherapy - Day 22: 0.5-1 hour postdose | 7.212 (55.84) | 5.370 (100.9) | 6.130 (144.9) | 5.350 (75.21) |  |  |
  Combination therapy - Day 15: Pre-dose: number analyzed (Participants) | 29 | 32 | 26 | 17 | 39 | 27 | 27
  Combination therapy - Day 15: Pre-dose | 1.848 (172.3) | 0.6526 (847.8) | 1.773 (92.68) | 1.744 (103.7) | 1.544 (102.3) | 1.400 (423.2) | 0.9718 (663.6)
  Combination therapy - Day 15: 0.5-1 hour postdose: number analyzed (Participants) | 26 | 31 | 26 | 15 | 39 | 27 | 26
  Combination therapy - Day 15: 0.5-1 hour postdose | 5.008 (74.54) | 2.805 (234.2) | 4.288 (136.4) | 3.226 (60.08) | 5.439 (70.73) | 5.922 (98.89) | 6.549 (72.47)
  Combination therapy - Day 15: 1-3 hour postdose: number analyzed (Participants) | 25 | 30 | 27 | 14 | 0 | 27 | 0
  Combination therapy - Day 15: 1-3 hour postdose | 8.038 (38.24) | 4.018 (155.6) | 5.897 (90.04) | 4.804 (57.38) |  | 7.644 (55.09) |
  Combination therapy - Day 15: 3-6 hour postdose: number analyzed (Participants) | 25 | 30 | 26 | 14 | 0 | 27 | 0
  Combination therapy - Day 15: 3-6 hour postdose | 7.811 (38.68) | 5.217 (51.57) | 6.322 (43.84) | 5.491 (35.36) |  | 5.717 (57.30) |
  Combination therapy - Day 15: 6-12 hour postdose: number analyzed (Participants) | 24 | 30 | 26 | 12 | 0 | 27 | 0
  Combination therapy - Day 15: 6-12 hour postdose | 5.186 (49.67) | 2.820 (60.56) | 3.661 (57.35) | 3.679 (52.80) |  | 3.023 (74.63) |

17. Secondary Outcome: Second Stage Cohort: Serum Concentrations of Bevacizumab
Description: Blood samples were collected to determine the serum concentration of bevacizumab.
Time Frame: Pre-dose and within 10 minutes of end of infusion on Days 1 and 85; Pre-dose on Days 29 and 169; and 90 days post last dose of bevacizumab. Assessed until DCO 17 Sep 2021
Population: The bevacizumab PK analysis set included all participants who received at least 1 dose of bevacizumab and provided any post-dose evaluable bevacizumab PK concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Second Stage: Ovarian Cancer Triplet
Number analyzed (Participants) | 31
mcg/mL
  Day 1: Pre-dose: number analyzed (Participants) | 25
  Day 1: Pre-dose | NA (NA) — NA = Below LLOQ. The LLOQ of bevacizumab is 0.5 mcg/mL.
  Day 1: End of infusion: number analyzed (Participants) | 28
  Day 1: End of infusion | 243.7 (30.01)
  Day 29: Pre-dose | 104.6 (29.30)
  Day 85: Pre-dose: number analyzed (Participants) | 26
  Day 85: Pre-dose | 145.5 (28.26)
  Day 85: End of infusion: number analyzed (Participants) | 21
  Day 85: End of infusion | 364.0 (23.74)
  Day 169: Pre-dose: number analyzed (Participants) | 25
  Day 169: Pre-dose | 147.9 (118.0)
  90 days post last dose: number analyzed (Participants) | 10
  90 days post last dose | 5.094 (224.1)

18. Secondary Outcome: Initial and Second Stage Cohorts: Number of Participants With Anti-Drug Antibody (ADA) Response to MEDI4736
Description: Blood samples were measured for the presence of ADAs and ADA-neutralizing antibodies (nAb) for MEDI4736 using validated assays. ADA prevalence was defined as the percentage of participants with positive ADA result at any time, baseline or post-baseline. ADA incidence (treatment-emergent ADA) was defined as the sum of both treatment-induced (post-baseline ADA positive only) and treatment-boosted ADA. Treatment-boosted ADA was defined as baseline ADA titer that was boosted to 4-fold or higher following drug administration. Persistently positive was defined as positive at >=2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive.
Time Frame: Pre-dose on Days 1, 15, 57, 85, 113 and 169; and 90 days post-last dose of MEDI4736. Assessed until DCO 14 Jun 2019 and 17 Sep 2021 for initial and second stage cohorts, respectively
Population: The ADA analysis set included all participants in the safety analysis set who have non-missing baseline ADA and at least 1 non-missing post-baseline ADA result for MEDI4736.
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
Number analyzed (Participants) | 33 | 32 | 31 | 35 | 0 | 29 | 25
Participants
  ADA prevalence | 0 | 1 | 0 | 0 |  | 0 | 0
  ADA incidence | 0 | 0 | 0 | 0 |  | 0 | 0
  ADA positive post-baseline and positive at baseline | 0 | 0 | 0 | 0 |  | 0 | 0
  ADA positive post-baseline and not detected at baseline | 0 | 0 | 0 | 0 |  | 0 | 0
  ADA not detected post-baseline and positive at baseline | 0 | 0 | 0 | 0 |  | 0 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0 |  | 0 | 0
  Persistent positive | 0 | 0 | 0 | 0 |  | 0 | 0
  Transient positive | 0 | 0 | 0 | 0 |  | 0 | 0
  Any nAb positive among any ADA positive | 0 | 0 | 0 | 0 |  | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were reported from the first dose administration up to 90 days following the date of last dose of study treatment. Assessed until DCO 14 Jun 2019 for initial stage cohorts except for ovarian cancer cohort and DCO 17 Sep 2021 for initial stage ovarian cancer cohort and second stage cohorts.
Description: The safety analysis set included all participants who received at least 1 dose of study treatment.
  For initial stage cohorts except ovarian cancer cohort: MedDRA 22.0. For initial stage ovarian cancer and second stage cohorts: MedDRA 24.0.
Arm/Group | Initial Stage: Small Cell Lung Cancer | Initial Stage: Breast Cancer | Initial Stage: Ovarian Cancer | Initial Stage: Gastric Cancer | Second Stage: Ovarian Cancer Expansion | Second Stage: Ovarian Cancer Triplet | Second Stage: Ovarian Cancer Doublet
All-Cause Mortality (participants affected / at risk) | 36/40 | 24/34 | 26/34 | 35/40 | 13/51 | 17/31 | 20/32
Serious Adverse Events (participants affected / at risk) | 23/40 | 4/34 | 10/34 | 10/40 | 13/51 | 6/31 | 8/32
Other Adverse Events (participants affected / at risk) | 40/40 | 34/34 | 32/34 | 40/40 | 50/51 | 31/31 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Stage: Small Cell Lung Cancer (N=40) | Initial Stage: Breast Cancer (N=34) | Initial Stage: Ovarian Cancer (N=34) | Initial Stage: Gastric Cancer (N=40) | Second Stage: Ovarian Cancer Expansion (N=51) | Second Stage: Ovarian Cancer Triplet (N=31) | Second Stage: Ovarian Cancer Doublet (N=32)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Stage: Small Cell Lung Cancer (N=40) | Initial Stage: Breast Cancer (N=34) | Initial Stage: Ovarian Cancer (N=34) | Initial Stage: Gastric Cancer (N=40) | Second Stage: Ovarian Cancer Expansion (N=51) | Second Stage: Ovarian Cancer Triplet (N=31) | Second Stage: Ovarian Cancer Doublet (N=32)
Non-cardiac chest pain (General disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 29 (33) | 14 (28) | 19 (55) | 15 (18) | 25 (39) | 18 (41) | 13 (20)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 2 (4) | 1 (1) | 2 (2) | 4 (8) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 4 (9) | 0 (0) | 8 (14) | 9 (12) | 5 (6)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 5 (5) | 5 (10) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (4) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 3 (3)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 5 (7) | 0 (0) | 5 (5) | 5 (5) | 1 (1) | 3 (4) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 4 (5) | 1 (1) | 3 (5) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 5 (5) | 6 (6) | 0 (0) | 10 (11) | 2 (2) | 5 (5)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 14 (15) | 10 (13) | 11 (14) | 16 (22) | 21 (23) | 8 (8) | 8 (9)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 5 (6) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 5 (6) | 7 (7) | 1 (1) | 3 (3) | 4 (5) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 18 (26) | 20 (27) | 26 (56) | 20 (24) | 34 (51) | 23 (44) | 28 (46)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 3 (4) | 5 (13) | 2 (2) | 8 (8) | 7 (8) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (18) | 11 (12) | 14 (39) | 17 (28) | 20 (37) | 16 (27) | 4 (6)
Asthenia (General disorders) | 7 (8) | 8 (8) | 2 (3) | 5 (5) | 6 (6) | 1 (2) | 7 (8)
Early satiety (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 16 (18) | 22 (29) | 20 (28) | 11 (11) | 28 (36) | 16 (25) | 16 (22)
Neutropenia (Blood and lymphatic system disorders) | 2 (4) | 5 (8) | 3 (5) | 2 (2) | 4 (4) | 3 (8) | 4 (5)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (3)
Mucosal inflammation (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 6 (7) | 1 (1) | 4 (7) | 5 (5) | 1 (1) | 3 (3) | 4 (5)
Pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Bronchitis (Infections and infestations) | 4 (6) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 2 (4) | 2 (2)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 2 (6) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (6) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (4) | 5 (6) | 1 (1) | 6 (6) | 2 (2) | 3 (3)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 3 (7)
Amylase increased (Investigations) | 4 (4) | 0 (0) | 5 (6) | 3 (3) | 2 (2) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (4) | 2 (2) | 1 (1) | 8 (15) | 7 (12) | 2 (2)
Blood creatinine increased (Investigations) | 8 (10) | 3 (4) | 1 (2) | 1 (1) | 6 (10) | 5 (11) | 7 (11)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 3 (5) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (2) | 4 (16) | 2 (2) | 0 (0) | 3 (5) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 4 (5) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 4 (4)
Platelet count decreased (Investigations) | 5 (5) | 2 (2) | 3 (27) | 1 (1) | 0 (0) | 4 (7) | 1 (1)
Thyroid function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 6 (7) | 3 (3) | 8 (9) | 14 (16) | 12 (14) | 7 (8) | 3 (3)
Weight increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
White blood cell count decreased (Investigations) | 5 (8) | 6 (21) | 4 (9) | 0 (0) | 4 (9) | 4 (6) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 14 (17) | 5 (6) | 10 (15) | 15 (15) | 10 (12) | 12 (19) | 9 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 2 (6) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (8) | 10 (12) | 2 (2) | 6 (8) | 9 (11) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (4) | 7 (12) | 2 (2) | 8 (8) | 5 (5) | 7 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 5 (6) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 1 (1) | 2 (2) | 5 (6) | 3 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 5 (6) | 4 (5) | 4 (4) | 5 (5) | 7 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 4 (5) | 2 (2) | 6 (6) | 3 (4) | 4 (5)
Disturbance in attention (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3) | 5 (5) | 6 (6) | 9 (12) | 3 (3) | 3 (3)
Dysgeusia (Nervous system disorders) | 3 (3) | 8 (8) | 5 (7) | 0 (0) | 7 (7) | 4 (5) | 6 (7)
Headache (Nervous system disorders) | 9 (10) | 7 (11) | 6 (10) | 4 (4) | 8 (11) | 11 (22) | 7 (9)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (1) | 2 (7) | 3 (5) | 2 (2) | 3 (3) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 6 (6) | 4 (4) | 1 (1) | 4 (4) | 3 (3) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5) | 4 (5) | 2 (2) | 8 (8) | 4 (4) | 5 (5)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 3 (3) | 3 (4) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (11) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 10 (15) | 5 (9) | 5 (5) | 11 (15) | 5 (5) | 3 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 5 (6) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 3 (4) | 11 (18) | 2 (2) | 13 (18) | 4 (6) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (9) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 3 (5) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 3 (4) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 10 (11) | 0 (0) | 3 (3) | 5 (7) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 6 (7) | 3 (5) | 6 (8) | 3 (4) | 5 (5)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5) | 9 (16) | 6 (9) | 7 (11) | 7 (10) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 5 (6) | 0 (0) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (6) | 8 (19) | 2 (4)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 2 (2) | 7 (8) | 1 (3) | 0 (0) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 6 (10) | 6 (9) | 8 (9) | 15 (19) | 8 (10) | 6 (9)
Abdominal pain upper (Gastrointestinal disorders) | 9 (12) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 12 (14) | 12 (20) | 11 (16) | 17 (28) | 12 (27) | 14 (21)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 7 (7) | 5 (5) | 6 (6) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 4 (4) | 3 (3) | 2 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT02734004/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT02734004/SAP_001.pdf